CLINICAL TRIAL: NCT02348775
Title: Glutathione and Function in HIV Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Rajagopal V Sekhar, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-34781 HIV-GSH
Record Dates: First submitted 2015-01-15; First posted 2015-01-28 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: HIV Infection; Erythrocyte Glutathione Deficiency
MeSH Terms: conditions — HIV Infections | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GlyNAC (Experimental): HIV infected subjects will be studied before and after taking oral glycine and n-acetylcysteine for 3 months
  Interventions: Dietary Supplement: GlyNAC (combination of glycine and n-acetylcysteine)

INTERVENTIONS:
Dietary Supplement: GlyNAC (combination of glycine and n-acetylcysteine) — HIV patients will be studied before and after receiving GlyNAC

SUMMARY:
We have recently reported that older patients with HIV are deficient in glutathione (GSH) due to decreased availability of cysteine and glycine, and that oral supplementation with cysteine (as n-acetylcysteine) and glycine for 2-weeks corrects their own levels, and improves (but does not fully normalize) concentrations of red-cell GSH. We also found that when GSH deficient, subjects had impaired mitochondrial fuel oxidation and this improved with an increase in intracellular GSH concentrations. These older HIV patients also had significant increases in muscle strength with improvement of GSH levels.The current proposal in older HIV patients will investigate study if cysteine and glycine supplementation for a duration of 12 weeks will result in changes in : (a) GSH levels; (b) body composition/anthropometry; (c) strength and function; (d) quality of life; (e) mitochondrial energetics; (f) biochemistry (including dyslipidemia and oxidative stress); (g) protein and glucose metabolism; (h) cognition and memory. After completing supplementation for 3 months, GSH concentrations, strength, function, mitochondrial energetics and neurocognitive tests will be measured for a further 2 months to determine the effects of washout.

DETAILED DESCRIPTION:
Detailed data are not as yet available

ELIGIBILITY:
Inclusion Criteria:

HIV patients:

* age 45-65 years

Non-HIV subjects:

* age 45-65 years

Exclusion Criteria:

1. Hospitalization in the past 3 months
2. Untreated hypothyroidism or hyperthyroidism
3. Known diabetes mellitus, hypercortisolemia, coronary artery disease.
4. Known liver impairment (ALT and AST >2ULN)
5. Renal impairment (Creatinine>1.4)
6. Inability to walk
7. Patients on anticoagulation or antiplatelet therapy.
8. Patient with triglyceride concentrations >500 mg/dl.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2018-12 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R V Sekhar, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor Metabolic Research Unit (MRU), Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will be submitted for publication once analyses are completed

RESULTS

PARTICIPANT FLOW:
Groups:
- GlyNAC: 8 HIV infected subjects were studied before and after receiving GlyNAC (combination of glycine and n-acetylcysteine) for 12-weeks
- Control Arm: This comprised of 8 participants not known to have HIV, and did not receive GlyNAC
Period: Overall Study
Arm/Group | GlyNAC | Control Arm
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cysteine/Glycine: 8 HIV infected subjects were studied before and after taking oral cysteine (as n-acetylcysteine) and glycine for 3 months, and compared to 8 uninfected controls
  Cysteine (as n-acetylcysteine) and glycine: Only HIV patients were studied before and after receiving cysteine and glycine
- No Supplements: 8 uninfected participants served as controls and were not supplemented
- Total: Total of all reporting groups
Arm/Group | Cysteine/Glycine | No Supplements | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (4.4) | 55 (3.6) | 55 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Muscle Glutathione Concentration
Description: Muscle glutathione concentrations measured by liquid chromatography
Time Frame: 20-weeks
Measure: Mean (Standard Deviation); unit: micromol/g.Hb
Groups:
- GlyNAC: 8 HIV infected subjects were studied before and after receiving oral GlyNAC (glycine plus n-acetylcysteine) for 12-weeks
Arm/Group | GlyNAC | Control Arm
Number analyzed (Participants) | 8 | 8
micromol/g.Hb | 0.5 (0.2) | 2.2 (0.8)

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- GlyNAC Arm: HIV infected subjects will be studied before and after taking GlyNAC for 12-weeks
- Control Arm: Controls will be HIV negative and not receive GlyNAC
Arm/Group | GlyNAC Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT02348775/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT02348775/SAP_001.pdf